CLINICAL TRIAL: NCT03457454
Title: Reducing Rural Colon Cancer Disparities Through Multi-level Interventions in Follow-up After Abnormal Screening Tests
Brief Title: Reducing Rural Colon Cancer Disparities
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201704046; U01CA209861-01A1 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Physicians, Primary Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary Care Provider/Staff Participants Interviews: * Up to two primary care providers and at least one staff person at each of the 16 clinics, with approximately 5 interviewees per clinic. Eligible providers and staff include physicians, nurse practitioners, nurses, case managers, medical assistants, administrative staff, or other employees of the clinic involved in the cancer screening and follow-up process.
  * If the participant verbally consents, the research team member will conduct an interview with the provider to learn about the current processes used to support and monitor colorectal cancer screening (CRC) from screening initiation through follow-up; assess capacity and interest in implementing Evidence Based Practices for supporting and monitoring CRC screening, including any ideas interviewees have or find appealing; and engage the organizations as partners to build interest, capacity, and infrastructure for future intervention trial and other future studies.
  Interventions: Other: Primary Care Provider/Staff Participants Interview
- Patient Participants Interviews: * 10 patients across 5 clinics will be recruited for interviews, which will address the patient experience with screening and follow-up.
  * If the participant verbally consents, the research team member will conduct an interview with the patient participant to gain a deeper understanding of the CRC screening process from the patient's perspective; the gaps, challenges, or road blocks/speed bumps to completing CRC screening steps; and what organizations can do better or differently to help people complete the CRC screening process.
  Interventions: Other: Patient Participant Interview
- Patient Participants Anonymous Survey: -Patient participants will be recruited to take an anonymous mailed survey, which will address patient level barriers to screening and follow-up focusing on out of pocket costs.
  Interventions: Other: Patient Participant Anonymous Survey
- Colonoscopy Provider/Staff Participants Interviews: * Colonoscopy providers and a staff or mid-level provider in each office will be recruited for interviews.
  * If the participant consents, the research team member will conduct an interview to learn about current processes used to support and monitor colorectal cancer screening from the perspective of gastroenterology/colonoscopy sites and to learn about how gastroenterology/colonoscopy sites communicate and coordinate care with other healthcare organizations and patients to support and monitor colorectal cancer screening.
  Interventions: Other: Colonoscopy Provider/Staff Participants Interviews

INTERVENTIONS:
Other: Primary Care Provider/Staff Participants Interview — -Approximately a 30 minute interview
  Groups: Primary Care Provider/Staff Participants Interviews
Other: Patient Participant Interview — -Approximately 45-60 minute interview
  Groups: Patient Participants Interviews
Other: Patient Participant Anonymous Survey — -Survey completion will take approximately 15 minutes
  Groups: Patient Participants Anonymous Survey
Other: Colonoscopy Provider/Staff Participants Interviews — -Approximately a 30 minute interview
  Groups: Colonoscopy Provider/Staff Participants Interviews

SUMMARY:
The investigators will conduct pre-implementations assessments of primary care clinics within a rural health system to determine current practices and capacities regarding colorectal cancer (CRC) screening and follow-up, preferred evidence-based interventions (EBIs) to improve follow-up, and factors that could influence successful implementation and eventual impact of a multi-level intervention to increase timely and complete follow-up after positive fecal occult blood test (FOBT) in rural patients.

ELIGIBILITY:
Inclusion Criteria for Primary Care Provider/Staff Participants -Eligible providers and staff include physicians, nurse practitioners, nurses, case managers, medical assistants, administrative staff, or other employees of the clinic involved in the cancer screening and follow-up process.

Inclusion Criteria for Patient Participants (Interview)

-Positive FOBT or colonoscopy

Inclusion Criteria for Patient Participants (Survey)

* 50 years of age or older
* Had a colonoscopy at one of Southern Illinois Healthcare's facilities within the last 24 months

Inclusion Criteria for Colonoscopy Provider/Staff Participants -Provider and a staff or mid-level provider in each office (5 colonoscopy providers in the Southern Illinois Healthcare region)

Exclusion Criteria for Primary Care Provider/Staff Participants

-None

Exclusion Criteria for Patient Participants (Interview)

* Negative FOBT or colonoscopy
* Exclusion Criteria for Patient Participants (Survey)
* Younger than 50 years of age

Exclusion Criteria for Colonoscopy Provider/Staff Participants None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Providers/Staff Participants, Patient Participants, and Colonoscopy Provider/Staff Participants from Southern Illinois Healthcare.
Sampling Method: Non-Probability Sample
Enrollment: 431 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Determine current practice and capacity regarding screening and follow-up of colorectal cancer screening at rural health clinics | Through completion of study (estimated to be 18 months)
  -This will be measured by interviews
Assess factors that could influence implementation of multi-level EBIs | Through completion of study (estimated to be 18 months)
  -This will be measured by interviews
Evaluate the capacity for colonoscopy and diagnostic follow-up by identifying those clinics/practitioners who deliver colonoscopy | Through completion of study (estimated to be 18 months)
  -This will be measured by interviews
Assess the care coordination and communication with primary care providers by colonoscopy clinics/practitioners | Through completion of study (estimated to be 18 months)
  -This will be measured by interviews

CONTACTS AND LOCATIONS:
Overall Officials: Aimee James, Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Southern Illinois Healthcare, Carbondale, Illinois
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu